CLINICAL TRIAL: NCT06515600
Title: Does Flow Trigger Sensitivity Adjustment Is Translational Mechanisms For Therapeutically Alternatives In Ventilator-Induced Diaphragm Dysfunction Critically Ill Patients?
Brief Title: Therapeutically Alternatives In Ventilator-Induced Diaphragm Dysfunction Critically Ill Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ibrahim Abuzaid, Director, Head of Department of Physiotherapy for Cardiovascular/Respiratory and Geriatrics, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Diaphragm Dysfunction
Record Dates: First submitted 2024-06-19; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Ventilator-Induced Diaphragmatic Dysfunction
Keywords: Trigger Sensitivity; Diaphragmatic dysfunction; Mechanical Ventilator; Minute Ventilation; Tidal Volume

STUDY DESIGN:
Intervention Model Description: Our Study was performed on sixty patients with VIDD from both genders. All patients will be referred by a physician. All patients were randomly assigned into two groups equal in number
Who Masked: Participant
Masking Description: Our Study was performed on sixty patients with VIDD from both genders. All patients will be referred by a physician. All patients were randomly assigned into two groups equal in number
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Group (A) (study group) will include 30 patients who practiced flow trigger sensitivity adjustment on mechanical ventilation for 1 week twice daily in addition to their plan of treatment.
  Interventions: Device: Practice flow trigger sensitivity adjustment on mechanical ventilation for 1 week twice daily in addition to their plan of treatment.
- Controlled group (Active Comparator): Group (B) (controlled group) will include 30 patients who received their routine plan of weaning of mechanical ventilator (controlled mode then spontaneous mode and finally spontaneous breathing trial).
  Interventions: Device: Practice flow trigger sensitivity adjustment on mechanical ventilation for 1 week twice daily in addition to their plan of treatment.

INTERVENTIONS:
Device: Practice flow trigger sensitivity adjustment on mechanical ventilation for 1 week twice daily in addition to their plan of treatment. — All patients were investigated by routine investigation (vital signs, arterial blood gas, ventilator mode, and the parameters).
  Two sessions were implemented per day for the study group for one week. The Trigger sensitivity adjustment trial begins with applying a load of 30% of the first recorded Negative Inspiratory Force (NIF).
  1. st Day 1st session, 30% 5 min.
  2. nd session, 30% 10 min.
  2nd Day 1st session, 30% 15 min 2nd session, 30% 20 min.
  3rd Day 1st session, 30% 25 min. 2nd session, 30% 30 min.
  4th Day 1st session, 40% 5 min. 2nd session, 40% 10 min.
  5th Day 1st session 40% 15 min 2nd session 40% 20 min.
  6th Day 1st session 40% 25 min. 2nd session 40% 30 min.
  7th Day 1st session 50% 5 min. 2nd session 50% 10 min.

SUMMARY:
The study is a prospective experimental study on adult patients admitted to the Critical Care Department in Qasr Al-Ainy. This study is conducted prospectively to assess the efficiency of trigger sensitivity adjustment on patients with ventilator-induced diaphragmatic dysfunction (VIDD).

DETAILED DESCRIPTION:
The study is a prospective experimental study on adult patients admitted to the Critical Care Department in Qasr Al-Ainy. This study is conducted prospectively to assess the efficiency of trigger sensitivity adjustment on patients with ventilator-induced diaphragmatic dysfunction (VIDD).1. Flow Trigger: This type of trigger responds to the gas flow during inspiration. A flow trigger measures the rate of change of flow as the patient begins to inhale. When the flow reaches a certain threshold, the ventilator is triggered to deliver a breath.

1. Laboratory investigations: Arterial blood gases (ABG):- (PH, PCO2, HCO3, and PO2) after the session.
2. Ventilator Parameters:( a) Minute Ventilation, b) Tidal Volume, c) Rapid Shallow breathing index, d) Negative Inspiratory Force (NIF) will be measured pre and post-treatment

ELIGIBILITY:
Age (years)

Weight (kg)

Height (cm)

BMI (kg/m²)

Inclusion Criteria:

* Patients who had undergone MV for 48 hours or more in a controlled mode.
* Patients could not generate maximum inspiratory pressure of more than 15 mbar
* Patients had diaphragmatic excursion less than 3 cm. (normal level from 3 to 5 cm.)(It can increase in a condition person to 7-8 cm).
* Patients had a diaphragmatic thickness fraction of less than 30%

Exclusion Criteria:

* Patients with comorbidities interfering and compromising weaning like cardiac arrhythmia, pericardial effusion, congestive heart failure, or unstable acute coronary syndrome.
* Patients who had inadequate training performance of the inspiratory muscle such as those having myopathy or neuropathy.
* Patients hemodynamically unstable.
* Patients who had a major neurological deficit.
* Sedated Patients.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Vital signs | one week
  Heart Rate (HR) b/min
Respiratory rate RR/min | one week
  Respiratory rate RR/min
Blood Pressure mmHg | one week
  Blood Pressure mmHg
Arterial blood gases (ABG):- | one week
  PH
PCO2 mmHg | one week
  PCO2 mmHg
HCO3 mEQ/Liter | one week
  HCO3 mEQ/Liter
PSAO2 mmHg | one week
  PSAO2 mmHg

SECONDARY OUTCOMES:
Ventilator parameters | one week
  Minute Ventilation L/min
Tidal Volume L/breath | one week
  Tidal Volume L/breath

IPD SHARING:
Plan to Share IPD: No
After publication

REFERENCES:
- [Result] Penuelas O, Keough E, Lopez-Rodriguez L, Carriedo D, Goncalves G, Barreiro E, Lorente JA. Ventilator-induced diaphragm dysfunction: translational mechanisms lead to therapeutical alternatives in the critically ill. Intensive Care Med Exp. 2019 Jul 25;7(Suppl 1):48. doi: 10.1186/s40635-019-0259-9. PMID 31346802
- [Result] Esteban A, Ferguson ND, Meade MO, Frutos-Vivar F, Apezteguia C, Brochard L, Raymondos K, Nin N, Hurtado J, Tomicic V, Gonzalez M, Elizalde J, Nightingale P, Abroug F, Pelosi P, Arabi Y, Moreno R, Jibaja M, D'Empaire G, Sandi F, Matamis D, Montanez AM, Anzueto A; VENTILA Group. Evolution of mechanical ventilation in response to clinical research. Am J Respir Crit Care Med. 2008 Jan 15;177(2):170-7. doi: 10.1164/rccm.200706-893OC. Epub 2007 Oct 25. PMID 17962636